CLINICAL TRIAL: NCT01224509
Title: Cervical Prostaglandin EP3 Receptor mRNA Expression 48 Hours After Administration of Mifepristone
Brief Title: The Effect of Mifepristone on the Expression of Cervical Prostaglandin EP3 Receptors
Acronym: EP3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Longer than expected recruitment period.
Sponsor: University of Southern California (Other)
Responsible Party: Marie-Soleil Wagner, MD, University of Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EP3 receptors
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Cervical Prostaglandin EP3 Receptors; Pregnancy
Keywords: Cervix; EP3 receptors; Mifepristone; Prostaglandin; Receptors; Steroids
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Experimental)
  Interventions: Drug: Mifepristone
- Non-treatment (Active Comparator)
  Interventions: Other: Non-treatment

INTERVENTIONS:
Drug: Mifepristone — Administration of 200 mg of mifepristone orally 48 hours prior to a cervical biopsy and evacuation by dilatation and curettage of the endometrial cavity
  Other Names: mifeprex
  Arms: Mifepristone
Other: Non-treatment — Non-treatment prior to a cervical biopsy and evacuation by dilatation and curettage of the endometrial cavity
  Arms: Non-treatment

SUMMARY:
The purpose of this study is to determine the effect of mifepristone on the expression of three cervical EP3 receptor isoforms (EP3-2, EP3-3 and EP3-6) in pregnant women ≤63 days gestational age.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* ≥18 years old
* seeking termination of a viable intrauterine pregnancy of ≤63 days, without any evidence of a threatened or spontaneous abortion

Exclusion Criteria:

* medical problems
* confirmed or suspected ectopic pregnancy
* having taken medications in the seven days prior to enrollment that would affect PG synthesis or metabolism of mifepristone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The amount of expression of EP3 receptor mRNA levels in cervical tissue after the administration of mifepristone | 48 hours after the administration of mifepristone

SECONDARY OUTCOMES:
The degree of cervical dilation after the administration of mifepristone | 48 hours after the administration of mifepristone

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Soleil Wagner, MD, Principal Investigator — University of Southern California; John K Jain, MD, Principal Investigator — University of Southern California
Locations (1):
- Women's and Children's Hospital, Reproductive Research Center, Los Angeles, California, United States